CLINICAL TRIAL: NCT00006151
Title: Combining a Smoke Ending Aid With Behavioral Treatment
Brief Title: Combining a Smoke Ending Aid With Behavioral Treatment - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Gariti (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Peter Gariti, Sponsor-Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-11645-1; R01DA011645 (NIH)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine fading; Accu Drop; cigarette tapering; smoking cessation; motivational interviewing
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accu Drops (AD&C) (Experimental): The experimental group (N=30) will be prescribed active Accu Drops (AD&C) plus behavioral therapy.
  Interventions: Behavioral: Behavioral Therapy
- Placebo (Placebo Comparator): The control condition (N=30) will be prescribed placebo Accu Drops (PD&C) plus behavioral therapy.
  Interventions: Behavioral: Behavioral Therapy

INTERVENTIONS:
Behavioral: Behavioral Therapy — Weekly behavioral therapy based on Project Match Motivational Therapy clinical manual plus systematic cigarette tapering.

SUMMARY:
The purpose of this study is to combine a smoke ending aid with behavioral treatment.

DETAILED DESCRIPTION:
The prime objective of this Innovative Stage I A/B Behavioral Therapy Development Research project is to conduct a pilot study under randomized, double-blind, placebo controlled conditions, to provide preliminary estimation of the efficacy of a 6 week Accu Drop nicotine fading protocol used in conjunction with cigarette tapering to bring about termination of cigarette usage in moderate to heavy smokers (*15 cpd) who are interested in smoking cessation. Both the experimental and control groups in this study will receive six weeks of the manually driven behavioral treatment by experienced and trained therapists. The experimental group (N=30) will also be prescribed active Accu Drops (AD&C) while the control condition (N=30) will be prescribed placebo Accu Drops (PD&C) very similar in appearance, viscosity, and taste to active Accu Drops. Completion of the study protocol and smoking cessation rates at 1 week, 1 month, and 6 months post-treatment will be the prime measures of efficacy. The findings of this study will provide sufficient preliminary indication for the efficacy of the experimental treatment and its extended investigation in a Phase II study or for its nonefficacy.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older, and no greater than 65 years of age
* Medically stable
* Smoke at least 15 filtered cigarettes daily
* Motivated to quit smoking

Exclusion Criteria:

* Medically unstable
* Currently psychiatrically unstable (schizophrenia, unstable psychosis, untreated major depression, active substance abuse within the past 6 months)
* Pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1999-05; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Gariti, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Gariti P, Alterman AI, Lynch KG, Kampman K, Whittingham T. Adding a nicotine blocking agent to cigarette tapering. J Subst Abuse Treat. 2004 Jul;27(1):17-25. doi: 10.1016/j.jsat.2004.03.005. PMID 15223089

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to a university based center for the study of addictions in 2002.
Pre-assignment Details: The study used a real world design meaning that participants were randomized on the same day as their study eligibility evaluation.
Groups:
- Accu Drops (AD&C): The experimental group (N=30) will be prescribed active Accu Drops (AD&C)
- Placebo (PD&C): The control condition (N=30) will be prescribed placebo Accu Drops (PD&C)
Period: Overall Study
Arm/Group | Accu Drops (AD&C) | Placebo (PD&C)
Started | 30 | 30
Completed | 17 | 16
Not Completed | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Accu Drop Plus Counseling: Active product and systematic cigarette tapering plus counseling.
- Placebo Accu Drop Plus Counseling: Placebo product and systematic cigarette tapering plus counseling
- Total: Total of all reporting groups
Arm/Group | Accu Drop Plus Counseling | Placebo Accu Drop Plus Counseling | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.07 (11.4) | 43.50 (12) | 45.29 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Abstinence Rate
Description: The main outcome measures were rates of treatment completion and smoking abstinence. It was hypothesized that the nicotine blocking agent product would lead to higher treatment completion rates, higher abstinence rates, and fewer problems with withdrawal than the placebo group.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Accu Drop Plus Counseling | Placebo Accu Drop Plus Counseling
Number analyzed (Participants) | 30 | 30
participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Accu Drops (AD&C) | Placebo (PD&C)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No